CLINICAL TRIAL: NCT02894190
Title: Development and Validation of the Beliefs About Ventilation Questionnaire (BVQ)
Brief Title: Development and Validation of the BVQ
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_BVQ_01
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2018-01

CONDITIONS: Chronic Respiratory Disease
Keywords: Non Invasive Ventilation (NIV); Adherence; Beliefs; Development; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main aim of this study is the development of the Beliefs about Ventilation Questionnaire (BVQ).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Indication to Non Invasive Ventilation (NIV), in three slots: <4; >4 e <12; <12 hours
* Outpatients or Inpatients
* Obstructive or restrictive reparatory disorder
* Voluntary agreement to be involved in the Study

Exclusion Criteria:

* Psychiatric Disorder
* Glasgow Coma Scale (CGS) <14
* Pure Obstructive Sleep Apnea Syndrome (OSAS)
* Tracheostomy with Invasive Ventilation (TIV) o Invasive Ventilation (IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with obstructive or restrictive respiratory diseases
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in adherence NIV in COPD patients at 3, 6 and 12 months as measured by the Beliefs of Ventilation Questionnaire (BVQ) | Baseline + After 3, 6 and 12 months following the recruitment

SECONDARY OUTCOMES:
Feasibility and acceptability of the questionnaire (duration / missing data) | Baseline + After 3, 6 and 12 months following the recruitment
Reliability over time of the questionnaire | Baseline + After 3, 6 and 12 months following the recruitment
External construct validity (The World Health Organization Quality of Life (WHOQOL); hours of Non Invasive Ventilation (NIV) prescribed, effective and referred by patients) | Baseline + After 3, 6 and 12 months following the recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Maria Nascente, Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Campos JL, Jara-Palomares L, Munoz X, Bustamante V, Barreiro E. Lights and shadows of non-invasive mechanical ventilation for chronic obstructive pulmonary disease (COPD) exacerbations. Ann Thorac Med. 2015 Apr-Jun;10(2):87-93. doi: 10.4103/1817-1737.151440. PMID 25829958
- [Result] Ozyilmaz E, Ugurlu AO, Nava S. Timing of noninvasive ventilation failure: causes, risk factors, and potential remedies. BMC Pulm Med. 2014 Feb 13;14:19. doi: 10.1186/1471-2466-14-19. PMID 24520952
- [Result] van Boven JF, Chavannes NH, van der Molen T, Rutten-van Molken MP, Postma MJ, Vegter S. Clinical and economic impact of non-adherence in COPD: a systematic review. Respir Med. 2014 Jan;108(1):103-13. doi: 10.1016/j.rmed.2013.08.044. Epub 2013 Sep 11. PMID 24070566